CLINICAL TRIAL: NCT02792907
Title: "Sensor Controlled Compliance Evaluation of Compressive Elastic Stockings Treatment in Patients After Elective Foot and Ankle Surgery" A Prospective, Randomized and Controlled Cohort Study
Brief Title: Sensor Controlled Compliance Evaluation of Compressive Elastic Stockings
Acronym: SENSCOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W568
Record Dates: First submitted 2016-05-25; First posted 2016-06-08 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Disorder of Ankle Joint
Keywords: Foot Surgery; Compliance; Compressive Stockings
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compressive Stockings group (Experimental): Patients with compressive stockings at the operated foot for 4 weeks
  Interventions: Device: Compressive stocking
- No compressive stockings group (No Intervention): Patients with no compressive stockings at the operated foot

INTERVENTIONS:
Device: Compressive stocking — After hindfoot and middlefoot surgery the patients from the Intervention Group will be treated with compressive stockings the removal of the suture. That means from the end of week 2 until the end of week 6 after surgery.
  Additionally the patients wearing behaviour is monitored by a electronic sensor, which is implanted in the patient´s stocking.
  Arms: Compressive Stockings group

SUMMARY:
Compressive stockings ameliorate functional outcome and quality of life in patients after elective orthopedic foot and ankle surgery. In this randomized controlled trial the investigators want to analyze the effect of compressive stockings after foot and ankle surgery. Additionally the investigators want to evaluate the compliance of the compressive stockings Treatment. Therefore an electronic chip device is implanted into the compressive stockings to monitor wearing time.

DETAILED DESCRIPTION:
Pain and swelling are typical sequelae following surgical procedures at the foot and ankle. While it is known that compressive stockings treatment decreases swelling and improves overall ankle function and quality of life in patients after ankle fracture, the investigators hypothesize that compressive stockings could also ameliorate functional outcome and quality of life in patients after elective orthopedic foot and ankle surgery.

Reduced compliance in wearing compressive stockings after foot and ankle surgery might probably be a limiting factor of this postoperative adjuvant compressive therapy. Therefore the investigators want to evaluate patient´s compliance by using an electronic chip device to monitor wearing behavior.

All patients who will be operated on their feet and ankle are randomized and blindly assigned into either the compressive or control-group. Each group consists of 80 patients (160 patients in total). The compression group includes patients who receive postoperative compression stockings. The control group does not receive any stockings. Regular checks at 6 weeks and 12 weeks postoperatively will be performed in order to assess the following parameters:

1. Foot and Ankle Scores
2. Pain

2. Swelling of the foot and lower limb 3. Wearing compliance by electronically recorded wearing time.

The Information about the implanted sensor, which records the stockings wearing time will be given to the patients after the compressive stockings therapy (6 weeks), so that the patients are not influenced by the fact, that their wearing behaviour had been measured.

After this information, the patients decide if the sensor information may be evaluated by the study team or not.

ELIGIBILITY:
Inclusion criteria:

* all patients with a signed informed consent
* all patients, who underwent hindfoot and middlefoot surgery

Exclusion criteria:

* patients with a externe Fixateur.
* patients with contraindication for the use of compressive stockings
* patients with severe General disease (cancer, rheumatoider Arthritis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Wearing Compliance | 6 weeks postoperatively
  With a sensor the wearing time in hours/day is monitored. Patients will be informed about the sensor at the 6 week follow up. They will be asked if the study Team is allowed to read the monitored wearing time.

SECONDARY OUTCOMES:
Pain | 12 weeks postoperatively
  Pain assessed in a visual analog scale ranging from 0-10 (0= no pain, 10= worst pain)
worker´s compensation | 12 weeks postoperatively
  % of ability to work the peroperative performed occupation.
pain killer use | 12 weeks postoperatively
  How many pills per day the patients require for the pain after surgery.
AOFAS | 12 weeks postoperatively
  American Orthopedic Foot and Ankle Score
Swelling | 12 weeks postoperatively
  Foot and ankle swelling measured in cm at defined Areas of the foot and ankle

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wirth, Dr. med., Principal Investigator — Balgrist University Hospital
Locations (1):
- Universtiy Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No